CLINICAL TRIAL: NCT03581318
Title: Technical and Translational Development of Cardiovascular MRI (CMR)
Brief Title: Technical and Translational Development of Cardiovascular Magnetic Resonance (CMR) Imaging
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180118; 18-H-0118
Record Dates: First submitted 2018-07-03; First posted 2018-07-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09-16

CONDITIONS: Normal and Abnormal Cardiovascular Physiology
Keywords: Congenital Heart Defects; Heart Valve Diseases; Chest pain (angina); Heart Failure; Coronary Heart Disease; CABG; CARDIOMYOPATHY; Atherosclerosis; MRI Technology Improvement
MeSH Terms: conditions — Heart Defects, Congenital; Heart Valve Diseases; Chest Pain; Angina Pectoris; Heart Failure; Coronary Disease; Cardiomyopathies; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Assessing Gadolinium deposition within the brain in healthy and patient subjects: Both healthy subjects and patient subjects who have previously undergone MRI and received gadolinium.
- Child Patient or Healthy Child: Healthy children will be used as controls for children with cardiac disease. Child patient will undergo MRI scans.
- Healthy Volunteers: Subjects will be used as controls for adults with cardiac disease.
- Research Patients Cardiac and Non Cardiac: Adults with cardiac disease that will undergo MRI scans.

SUMMARY:
Background:

Magnetic resonance imaging (MRI) is an important non-invasive tool to study and diagnose cardiovascular disease. MRI scanners use strong magnetic fields and radio waves to create pictures of body organs. Researchers want to find better MRI methods and new ways of imaging cardiovascular disease and better understand normal and abnormal cardiovascular and brain function. Researchers are also interested in seeing if gadolinium, the commonly used MRI contrast agent, stays in the body long after the MRI was performed.

Objectives:

To develop new methods for imaging the heart and other organs of the body.

To describe cardiovascular diseases using newer MRI methods

To look at the relationship between cardiovascular disease and cardiovascular risk factors and other organ systems

To look for gadolinium deposits in the brain from prior exams.

Eligibility:

Healthy people and people with known or suspected cardiovascular disease ages 7 and older may be eligible for this study.

Researchers may be particularly interested in those who:

* Have suspected or known cardiovascular disease
* Were previously exposed to a gadolinium-based contrast agent,
* Need to have a heart MRI scheduled
* Need a test of the heart or other body part or will be undergoing a future cardiac catheterization

Design:

There are multiple arms to the study with optional components; therefore, there are multiple variations as to what an individual participant s experience may involve.

Participants will have an MRI scan lasting up to 2 hours. The scanner is a large hollow tube. During the scan, there may be loud knocking and buzzing sounds caused by the scanner. Participants will lie on a table that slides in and out of the tube. Their vital signs may be monitored.

Participants may have a test of heart electrical activity using wires connected to pads on the skin.

Participants may have blood drawn.

Participants may be injected with an MRI contrast agent through a plastic tube inserted in the arm.

DETAILED DESCRIPTION:
The purpose of this protocol is to develop and test new MRI techniques applicable to patients undergoing cardiovascular evaluation with the ultimate goal of translating the technical advances into improving clinical diagnosis and management of patients undergoing cardiovascular evaluation. Patients undergoing cardiovascular evaluation and healthy volunteers will be scanned under the protocol. We will evaluate new developments in non-contrast and contrast MRI of the heart and blood vessels and novel postprocessing methods.

The use of the newer sequences will be used to improve clinical imaging workflow and disease diagnosis. We hope to use this protocol to clearly describe cardiovascular disease and associated problems using novel MRI methods and follow certain subsets of patients with disease as part of a natural history process. Inter-related physiologic systems may be phenotyped by MRI with characterization of disease associations between different organ systems.

Additionally, information regarding gadolinium deposition of the brain will be gathered. The literature regarding deposition of gadolinium in the brain has a large void regarding information of prevalence of the phenomenon in healthy subjects. The National Institutes of Health has a large healthy subject pool who have participated in gadolinium contrast MRI studies. This pool of healthy subjects is not easily available at most clinical MRI centers, and thus, we are uniquely well-situated to be able to answer this outstanding question.

For all objectives, MRI studies will be conducted in the NIH MRI systems located at the NIH Clinical Center in Bethesda, Maryland. These procedures may involve the intravenous administration of commercially available MR contrast media and exercise or pharmacologic stress testing. Results will be used to evaluate the performance of various research pulse sequences, gradient coils, and radiofrequency receiver coils on human subjects and will provide essential ground work for specific patient protocols, both diagnostic and therapeutic.

ELIGIBILITY:
* INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:
* Age greater than or equal to 7 years
* Able to follow instructions and lie still in the MRI scanner
* Currently without known cardiovascular disease
* Able to provide informed consent in writing or provide guardian consent
* Willingness to cooperate with all study procedures and available for scheduled study events

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Important past or chronic medical illness such as major cardiovascular conditions like myocardial infarction, congenital heart disease, and known cardiomyopathy
* Conditions that are thought to make MRI unsafe (that will be determined by filling out a separate form) including:

  * Cardiac pacemaker or implantable defibrillator unless it is labeled safe or conditional for MRI
  * Cerebral aneurysm clip unless it is labeled safe for MRI
  * Neural stimulator (e.g. TENS-Unit) unless it is labeled safe for MRI
  * Any type of ear or cochlear implant unless it is labeled safe for MRI
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet unless cleared by plain x-ray as safe for MRI
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe or conditional for MRI
* eGFR < 60 mL/min/1.73m^2 using the 2021 CKD-EPI equation or equivalent and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications. Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents
* Pregnancy. When uncertain of pregnancy status, subjects will undergo serum or urine pregnancy testing within the 7 days prior to the examination. Among those subjects who will receive MRI contrast , subjects of child-bearing potential will under serum or urine pregnancy testing within 7 days of the day prior to examination. In addition, the subject will be asked if she may be pregnant prior to the performance of the MRI, even if the pregnancy test was negative within the past week. The pregnancy test will be repeated if she answers in the affirmative. Post-menopausal and surgically sterilized subjects are automatically exempt from this testing.
* If receiving contrast, children and breast feeding women (unless subject is willing to discard breast milk for 24 hours) are excluded
* Healthy volunteer children will not have contrast
* In a years time, healthy volunteers are not restricted as to the number of non-contrast MRI examinations they undergo, but they may not undergo more than two examinations involving gadolinium-based contrast agents (GBCA) and those exposures will be at least 18 hours (12 half-ives) apart.

INCLUSION CRITERIA FOR SUBJECTS WITH KNOWN OR SUSPECTED WITH HEART DISEASE:

* Age greater than or equal to 7 years
* Subjects with known or suspected cardiovascular disease
* Able to provide informed consent in writing or provide guardian consent
* Willingness to cooperate with all study procedures (including food restriction) and available for scheduled study events

EXCLUSION CRITERIA FOR SUBJECTS WITH KNOWN OR SUSPECTED HEART DISEASE:

* Conditions that are thought to make MRI unsafe (that will be determined by filling out a separate form) including:

  * Cardiac pacemaker or implantable defibrillator unless it is labeled safe or conditional for MRI
  * Cerebral aneurysm clip unless it is labeled safe for MRI
  * Neural stimulator (e.g. TENS-Unit) unless it is labeled safe for MRI
  * Any type of ear or cochlear implant unless it is labeled safe for MRI
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet unless cleared by plain x-ray as safe for MRI
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe or conditional for MRI
* Pregnancy. When uncertain of pregnancy status, subjects will undergo serum or urine pregnancy testing within the 7 days prior to the examination. Among those subjects who will receive MRI contrast , subjects of child-bearing potential will undergo serum or urine pregnancy testing 7 days prior to the examination. In addition, the subject will be asked if she may be pregnant prior to the performance of the MRI, even if the pregnancy test was negative within the past week. The pregnancy test will be repeated if she answers in the affirmative. Post-menopausal and surgically sterilized subjects are automatically exempt from this testing.
* Breast feeding (unless subject is willing to discard breast milk for 24 hours if receiving contrast)
* eGFR < 30 mL/min/1.73m^2 using the 2021 CKD-EPI equation or Community Practice Standard for Pediatric case or equivalent and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications. Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents
* Cardiorespiratory instability as determined by the enrolling clinician

INCLUSION CRITERIA FOR SUBJECTS WITH NON-CARDIAC DISEASE:

* Age greater than or equal to 7 years
* Able to provide informed consent in writing or provide guardian consent
* Willingness to cooperate with all study procedures (including food restriction) and available for scheduled study events
* Known or suspected brain, hematology, oncology, endocrine, pulmonary, or other non-cardiac disease.

EXCLUSION CRITERIA FOR SUBJECTS WITH NON- CARDIAC DISEASE:

* Conditions that are thought to make MRI unsafe (that will be determined by filling out a separate screening form) including:

  * Cardiac pacemaker or implantable defibrillator unless it is labeled safe or conditional for MRI
  * Cerebral aneurysm clip unless it is labeled safe for MRI
  * Neural stimulator (e.g. TENS-Unit) unless it is labeled safe for MRI
  * Any type of ear or cochlear implant unless it is labeled safe for MRI
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet unless cleared by plain x-ray as safe for MRI
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe or conditional for MRI
* Pregnancy. When uncertain of pregnancy status, subjects will undergo serum or urine pregnancy testing within the 7 days prior to examination. Among those subjects who will receive MRI contrast , subjects of childbearing potential will undergo serum or urine pregnancy testing on the day of the examination. In addition, the subject will be asked if she may be pregnant prior to the

performance of the MRI, even if the pregnancy test was negative within the past week. The pregnancy test will be repeated if she answers in the affirmative. Post-menopausal and surgically sterilized subjects are automatically exempt from this testing.

* Breast feeding in those subjects receiving contrast (unless subject is willing to discard breast milk for 24 hours
* eGFR < 30 mL/min/1.73m^2 using the 2021 CKD-EPI equation14 or equivalent and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications. Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents
* Cardiorespiratory instability or as determined by the enrolling clinician

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Translational development of MRI sequences | on going
  Possible comparison to other studies that subjects may have undergone. Descriptive MRI catalogue of multiple cardiovascular processes Follow-up of outcomes subsequent to the MRI scan in select subject groups Follow-up of changes in diagnosis following the MRI scan in select subject groups
Technical development of MRI sequences | on going
  Possible assessments include structure depictions, heart chamber volumes, blood flow velocity, image quality scores, pixelwise and segmental summary scores of parametric maps in the heart. Anatomical imaging may be assessed for non- cardiac applications. Contrast- to-noise, and signal-to-noise measurements may be performed. For novel sequences, comparisons to standard product sequences may be performed.
Evaluating the correlation | on going
  Measurements of cardiac chamber size and function, vascular reactivity and perfusion are among the parameters that may be followed with comparison to standard biomarkers of disease and clinical manifestations of disease. Neurologic vascular reactivity, blood volume, resting state connectivity, BOLD signal changes may be compared among healthy subjects, asymptomatic subjects with risk factors, and subjects with disease.
Assesment of Gad deposition in the brain | on going
  Assessment of non-contrast MRI findings that are consistent with gadolinium deposition.

CONTACTS AND LOCATIONS:
Overall Officials: W. Patricia Bandettini, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The study team will make a decision on this matter.

REFERENCES:
- [Derived] Bandettini WP, Shanbhag SM, Mancini C, Henry JL, Lowery M, Chen MY, Xue H, Kellman P, Campbell-Washburn AE. Evaluation of Myocardial Infarction by Cardiovascular Magnetic Resonance at 0.55-T Compared to 1.5-T. JACC Cardiovasc Imaging. 2021 Sep;14(9):1866-1868. doi: 10.1016/j.jcmg.2021.02.024. Epub 2021 May 19. No abstract available. PMID 34023254
- [Derived] Bandettini WP, Shanbhag SM, Mancini C, McGuirt DR, Kellman P, Xue H, Henry JL, Lowery M, Thein SL, Chen MY, Campbell-Washburn AE. A comparison of cine CMR imaging at 0.55 T and 1.5 T. J Cardiovasc Magn Reson. 2020 May 18;22(1):37. doi: 10.1186/s12968-020-00618-y. PMID 32423456
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-H-0118.html